CLINICAL TRIAL: NCT06498427
Title: A Quasi-experimental Longitudinal Study of Adolescents' Well-being in Community-based Treatment Versus in a Psychiatric Residential Treatment Facility (PRTF)
Brief Title: Adolescents' Well-being in Community-based Treatment Versus Residential Treatment
Status: Completed | Type: Observational
Sponsor: Outcome Referrals, Inc. (Industry)
Collaborators: The Duke Endowment (Other); Children's Hope Alliance (Unknown)
Responsible Party: Sponsor
Other Study IDs: WCG IRB Protocol #20211997
Record Dates: First submitted 2024-06-25; First posted 2024-07-12 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Adolescent Well-Being; Mental Disorders, Severe
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Child ACTT - Experimental: Excerpt from the Partners Child ACTT service definition in North Carolina (Revised 5-23-19):
  Program Requirements: Child ACTT (Assertive Community Treatment Team) is a team-based multi-disciplinary approach to serve children in their homes, kinships placements, foster homes ... The team will have daily meetings to prioritize activities, share information, and discuss individual members. The team will be available to respond 24/7 for crisis de-escalation and assessment, inclusive of availability by phone within 15 minutes and face to face within no more than 2 hours. This will include face-to-face assessment by a clinician, or nurse if this is determined to be needed for the individual. The psychiatric provider will be available minimally by phone 24/7 for consultation and treatment recommendations. The team will assess the overall needs of the family to ensure that all necessary treatment and supports are in place for entire family system.
- PRTF - Treatment as Usual: Psychiatric Residential Treatment Facilities (PRTFs) are non-hospital facilities intended to provide inpatient services to Medicaid-eligible individuals who are under the age of 21. A PRTF's mission is to either improve residents' condition or prevent further regression to ultimately remove the need for such services. PRTFs provide a range of comprehensive services intended to treat residents' psychiatric conditions under the supervision and direction of a psychiatrist. The core components in a PRTF program include at least weekly medication management, 24 hours nursing services, high staff-to-client ratio with awake staff during night hours, individual, group, and family therapy, intensive psychoeducation, behavioral model of care designed to teach new functional skills, and comprehensive assessments as needed.

SUMMARY:
This is a quasi-experimental longitudinal study to compare the outcomes of youth in Psychiatric Residential Treatment Facility (PRTF) compared to youth in the at-home Child-Focused Assertive Community Treatment Team [Child ACTT] program. The hypothesis is that Child ACTT will be associated with better outcomes and lower cost than PRTF among adolescents admitted to Child ACTT or PRTF.

DETAILED DESCRIPTION:
Psychiatric Residential Treatment Facility (PRTF) care is expensive, removes adolescents from their communities, and is not necessarily effective. Managed care organizations (MCO) are exploring other methods of providing intensive care at home. Several states (e.g., Maine, Minnesota, Florida) have initiated and maintained Youth -Assertiveness Community Treatment (ACT) programs that are adapted from the evidence-based adult ACTT model. Children's Hope Alliance (CHA) has been offering the Child-Focused Assertive Community Treatment Team [Child ACTT] Program as a service for potential clients since December 2019.

RECRUITMENT PROCEDURES

1. The MCO will send a letter to PRTF treatment providers to inform them about this study.
2. CHA and the PRTFs will inform the legal guardians of children who meet the inclusion criteria about a potential study opportunity.
3. If the legal guardian verbally consents to being contacted by Outcome Referrals, Inc. (ORI) about the study, CHA or PRTF will forward the contact information for the legal guardian of the eligible participant to ORI via an encrypted email.
4. ORI will contact the legal guardian to describe the study and review the eligibility criteria with potential participants (within 5 days of treatment authorization).

Individuals who meet the eligibility criteria and are interested in participating in the study will be sent electronic copies of the assent and consent forms to review and sign. ORI will inform the original referral source (CHA or specific PRTF) if family is not able to be contacted or does not consent for study.

METHODS AND PROCEDURES

A randomized controlled trial was originally selected as the study design for this project because it is the gold standard for testing for causality; however, given recruitment issues, it was decided to transition to a quasi-experimental study instead. Although the investigators cannot conclude that one treatment is more efficacious than another, this quasi-experimental longitudinal study will provide important comparative information about these two treatment options for high need youth and families.

After study assent and consent forms are received by ORI, ORI will inform the referral source (CHA or PRTF) that the family consented to participate in the study: CHA or the PRTF will provide ORI with the contact information for the case manager at the facility for each participant. ORI will send an email to the case manager to inform them of that client's participation and request a time to train them on study assessment procedures.

ORI will administer a) the electronic assents and consents through an e-signature platform, and b) study assessments to both participants and their legal guardians during and post-treatment through ORI's secure platform, WellnessCheck.net.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages 12 and 18
* Has primary mental health diagnosis
* Admitted for treatment in a participating program (i.e., Psychiatric Residential Treatment Facility (PRTF) or Child ACTT)
* A trained ORI staff member determines that the youth is able to understand and sign an assent for participation
* Documentation of the youth's assent to participate in the study
* A legal guardian provides consent for the youth to participate in the study

Exclusion Criteria:

* The client is not admitted to treatment in a participating program
* The client has dropped out of this study during a previous treatment episode
* Client does not initiate treatment

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be recruited from PRTF and Child ACTT. For example, at Partners MCO in 2020, 131 unique members were served in PRTFs. Their summary demographic characteristics for gender, race, and age were as follows: 43.5 percent female and 55.7 percent male; 18 percent Black, 78 percent White, 3 percent Other and an average age of 14.5 years. Potential primary diagnoses expected are major depressive disorders, psychotic disorders, anxiety disorders, disruptive behavior disorders and bipolar disorder.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Mean change on average z-scores from participant self report on Clinical Scale of the Treatment Outcome Package (TOP-CS) over time | Baseline completed within 3 weeks of treatment start then a TOP every month up to Month 6 during treatment then at 3 months post-discharge.
  TOP is a comprehensive well-being assessment that is used in behavioral health and child welfare settings. The Adolescent TOP Clinical Scale (TOP-CS) is a 58-item scale for adolescents who are between the ages of 11 - 21. The TOP-CS assesses the client's past 2-week experience on 12 domains including Depression, Attention Problems, Conduct Disorders, and Suicidality (scores are risk-adjusted for case mix variables assessed via 37 items on the companion TOP-Case Mix form, such as divorce, job loss, comorbidity). Participants indicate "All" to "None of the Time" for each item on a 6-point Likert scale. The z-scores (standard deviation units relative to the general population mean for each domain) will be averaged together to create one summary score. Higher scores suggest higher severity/lower behavioral well-being.

SECONDARY OUTCOMES:
Satisfaction score most proximal to discharge (up to Month 6) from participant self report on the Overall Provider Quality subscale of the TOP Satisfaction Scale | Every month up to Month 6 during treatment
  The Overall Provider Quality subscale of the TOP Satisfaction Scale assesses patient satisfaction with behavioral health care. 4 Likert scale items about satisfaction with treatment plus single qualitative item (i.e., What are two reasons for your rating of the overall quality of the treatment received?). Scores range between 1 and 6 (higher scores indicate higher satisfaction).
Mean change on average z-scores from legal guardian ratings for the participants on the Treatment Outcome Package | Baseline completed within 3 weeks of treatment start then a TOP every month up to Month 6 during treatment then at 3 months post-discharge.
  See Outcome 1 description
Satisfaction score most proximal to discharge (up to Month 6) from legal guardian report on the Overall Provider Quality subscale of the TOP Satisfaction Scale | Every month up to Month 6 during treatment
  See Outcome 2 description
Mean change on the z-score for individual domains from participant self report on the Treatment Outcome Package | Baseline completed within 3 weeks of treatment start then a TOP every month up to Month 6 during treatment then at 3 months post-discharge.
  See Outcome 1 description

OTHER OUTCOMES:
Cost of treatment | Through study treatment completion, a maximum of 6 months
  Estimated treatment cost per condition will be assessed by calculating the number of days in treatment times cost per day

CONTACTS AND LOCATIONS:
Locations (1):
- Outcome Referrals, Inc., Framingham, Massachusetts, United States

REFERENCES:
- [Background] Kraus DR, Seligman DA, Jordan JR. Validation of a behavioral health treatment outcome and assessment tool designed for naturalistic settings: The Treatment Outcome Package. J Clin Psychol. 2005 Mar;61(3):285-314. doi: 10.1002/jclp.20084. PMID 15546147
- [Background] Baxter EE, Alexander PC, Kraus DR, Bentley JH, Boswell JF, Castonguay LG. Concurrent validation of the child and adolescent versions of the Treatment Outcome Package (TOP). Journal of Child and Family Studies. 2016; 25(8): 2415-2422.